CLINICAL TRIAL: NCT07318194
Title: Surgical Field Quality Assessment and Complications in Distal Radius Fractures Using the Minimum Inflation Tourniquet Pressure: Limb Occlusion Pressure Versus Arterial Occlusion Pressure. And Clinical, Radiological and Quality of Life Assessment at One-year Follow up. A Randomized Controlled Trial.
Brief Title: Surgical Field Quality Assessment and Complications in Distal Radius Fractures Using the Minimum Inflation Tourniquet Pressure.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari de Terrassa (Other)
Responsible Party: Principal Investigator, Josep Maria Mora Guix, MD, PhD. Chief of Shoulder Unit, Consorci Sanitari de Terrassa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01-23-105-045
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-05

CONDITIONS: Distal Radius Fracture
Keywords: Ischaemia; Arterial Occlusion Pressure; Limb Occlusion Pressure; Surgical field; Distal radius fracture
MeSH Terms: conditions — Wrist Fractures; Ischemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNEUMATIC TOURNIQUET USING LIMB OCCLUSION PRESSURE (Experimental): A distal sensor connected to the pneumatic tourniquet system is placed on the patient's index finger and automatically calculates the minimum ischaemia pressure required to occlude the distal blood flow.
  Interventions: Procedure: PNEUMATIC TOURNIQUET INFLATION PRESSURE
- PNEUMATIC TOURNIQUET USING ARTERIAL OCCLUSION PRESSURE (Active Comparator): Pneumatic cuff pressure is calculated by adding 100 mmHg to the patient's systolic blood pressure.
  Interventions: Procedure: PNEUMATIC TOURNIQUET INFLATION PRESSURE

INTERVENTIONS:
Procedure: PNEUMATIC TOURNIQUET INFLATION PRESSURE — Patients undergoing osteosynthesis of distal radius fractures will be randomised in two groups: pneumatic cuff pressure calculated based on Limb Occlusion Pressure, and pneumatic cuff pressure calculated based on Arterial Occlusion Pressure, without adding any security margin in any group.

SUMMARY:
Analyse surgical field bleeding, surgical time, and intraoperative pain in patients undergoing osteosynthesis of distal radius fractures using ischaemia pressure calculated based on Limb Occlusion Pressure, compared with Arterial Occlusion Pressure. Additionally, compare muscle damage and postoperative complications, and clinical, functional, quality of life and radiological outcomes at one-year follow-up.

DETAILED DESCRIPTION:
Randomised controlled clinical trial. It will be conducted with patients undergoing osteosynthesis of distal radius fractures (ischaemia pressure calculated according to Arterial Occlusion Pressure or Limb Occlusion Pressure), included consecutively at Terrassa Hospital from June 2023 to October 2025. The estimated sample size will be 70 patients per group. Pneumatic cuff pressure, ischaemia time, intraoperative ischaemia-related pain, surgical field bleeding, muscle damage, and postoperative complications will be assessed. One-year follow-up will include clinical, functional, quality-of-life, and radiological evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older, diagnosed with a distal radius fracture meeting surgical criteria.
* Surgery performed by the Hand Unit at Terrassa University Hospital.
* Axillary block as the anaesthetic technique.
* The surgeon completes all required study procedures.
* Written informed consent obtained from the patient.

Exclusion Criteria:

* Bilateral distal radius fractures.
* Osteosynthesis of an ipsilateral distal ulnar fracture.
* Requirement for general anaesthesia.
* High anaesthetic risk (ASA IV).
* Body mass index (BMI) > 40.
* Uncontrolled hypertension or treatment with more than three antihypertensive medications.
* Contraindications to tourniquet use, such as arteriovenous fistulas or peripheral vascular disease.
* Failure of the surgeon to complete the required study procedures.
* Lack of informed consent for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
SURGICAL FIELD BLEEDING | At the end of the surgery.
  Fromme scale (0-5). Assessed by the main surgeon. 0 (the best) - 5 (the worst)
ISCHAEMIA TIME | Measured at the end of the surgery.
  Measured in minutes. It refers to the duration from the onset of pneumatic ischemia until its cessation, prior to wound closure at the end of the surgery.
INTRAOPERATORY PAIN | Measured 60 minutes after the start of the surgery.
  Pain caused by the pneumatic cuff on the arm, measured using the Visual Analogue Scale (0-10).
  0 (the best) - 10 (the worst)
COMPLICATIONS | During the surgery or the immediate postoperative period.
  Any cutaneous, muscular, vascular or nervous complication.
MUSCLE DAMAGE | In postoperative blood tests 60 minutes after surgery.
  Assessed based on creatine kinase (CK) levels. Expressed in μmol/L.
LIMB OCCLUSION PRESSURE | Measured inside the operating room immediately prior to the start of surgery.
  Measured in mmHg. Automatically recorded by placing a distal sensor on the index finger (second digit) of the hand, connected to the pneumatic ischemia device. No safety margin will be applied. A single measurement will be taken.
ARTERIAL OCCLUSION PRESSURE | Measured inside the operating room immediately prior to the start of surgery.
  Expressed in mmHg. Calculated using the formula: systolic blood pressure + 100 mmHg.

SECONDARY OUTCOMES:
FRACTURE TYPE | Preoperative
  Measured in the wrist X-Ray using Frykman Scale (1-8).
SYSTOLIC BLOOD PRESSURE | Measured inside the operating room, after the patient has been lightly sedated.
  Expressed in mmHg. Measured in the limb to be treated.
PRWE TEST | Assessed one year postoperatively
  15-item questionnaire scoring pain and function (0-100 scale, 0=best/no problem, 100=worst)
QUICK-DASH TEST | Assessed one year postoperatively
  functionality scale. calculating a score from 0-100 where higher means more difficulty/worse function
RANGE OF MOVEMENT | Assessed one year postoperatively
  In degrees. Using a goniometer. Wrist flexion, extension, radial deviation, ulnar deviation, pronation supination.
GRIP STRENGTH | Assessed one year postoperatively.
  Expressed in kg. Using a dynamometer.
EUROQOL-5D TEST | Assessed one year postoperatively.
  Quality of life scale. The EQ-5D (EuroQol 5-Dimension) is a widely used questionnaire assessing health-related quality of life through five dimensions: Mobility, Self-care, Usual Activities, Pain/Discomfort, and Anxiety/Depression, each rated on a scale (3 or 5 levels).
SF-12 TEST | Assessed one year postoperatively.
  Quality of life scale. Scores above 50 indicate a better-than-average health-related quality of life. Scores below 50 suggest below-average health
BODY MASS INDEX | Preoperative
  Calculated according to weight (in kg) and height (in centimeters).
ARM CIRCUMFERENCE | Preoperative.
  Expressed in centimeters. Measured with a tape measure.

CONTACTS AND LOCATIONS:
Locations (1):
- JM Mora, Terrassa, Barcelona, 08227, Terrassa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided